CLINICAL TRIAL: NCT01383798
Title: How Does Iron Deficiency Without Anemia (IDNA) Affect Endurance Training In Female Collegiate Endurance Athletes?
Brief Title: How Does Iron Supplementation Affect Training and Performance in Female Collegiate Rowers?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OSP 57149
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-03

CONDITIONS: Iron Deficiency (Without Anemia)
Keywords: iron deficiency, physical performance, female athletes
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Red capsule (50 mg) lactose
  Interventions: Dietary Supplement: Placebo
- Ferrous sulfate (Experimental)
  Interventions: Dietary Supplement: Ferrous sulfate

INTERVENTIONS:
Dietary Supplement: Placebo — 100 mg lactose per day for 6 weeks
  Arms: Placebo
Dietary Supplement: Ferrous sulfate — 100 mg per day of ferrous sulfate for 6 weeks
  Arms: Ferrous sulfate

SUMMARY:
The specific aims of the current study were: 1) To determine the prevalence of IDNA in a sample of female rowers at the beginning of a training season; 2) To determine how IDNA affects endurance training and performance at the beginning of a training season; 3) To determine how iron supplementation affects iron status, training and performance in IDNA female collegiate rowers. The researchers hypothesized that IDNA affects endurance performance in female collegiate rowers both in and outside of the laboratory, and that iron supplementation of IDNA rowers will improve iron status, and consequently, training quality via increased energetic efficiency.

DETAILED DESCRIPTION:
Iron deficiency (ID) is the most common nutrient deficiency in the United States, affecting 13% of pre-menopausal women, and approximately 30% of physically-active women (1, 2). Iron deficiency anemia (IDA) is clinically defined as hemoglobin (Hgb) less than 12.0 g/dl. Iron depletion without anemia (IDNA), or low iron stores, is defined as Hgb greater than 12.0 g/dl and serum ferritin (sFer) less than 20.0 µg/L. Female athletes are at higher risk of IDNA due to their menstrual status, poor dietary intake, and high training volume and intensity (3). Consequences of IDNA that may be relevant to athletes include reduced work capacity, endurance, and energetic efficiency (4-6); and increased local muscle fatigue (7). The mechanism by which IDNA affects endurance and physical performance remains unclear, and the functional consequences of IDNA are not fully understood in trained individuals, as studies to examine these relationships have been underpowered (8, 9).

Our lab has previously reported the effects of iron deficiency on physical performance in untrained, IDNA women adapting to an aerobic training program. Hinton et al (5) showed that the effect of iron supplementation on physical performance was mediated by changes in iron status (sFer), and concluded that IDNA reduces the potential benefits of aerobic training on endurance. In that study, subjects who were supplemented with iron for 6 weeks during aerobic training improved their time to complete a 15-km cycling time trial by 3.4 min compared to 1.6 min in the placebo group (p<0.05). Given these convincing results, the study of highly-trained competitive female athletes training at a high volume and intensity was warranted. We expected these significant effects to persist in competitive collegiate athletes. However, we expected the magnitude of these effects to be somewhat less due to collegiate athletes' advanced training status, and thus a smaller margin of improvement in performance due to response of increased body iron stores. The goal of the proposed study was to determine whether marginal iron deficiency (IDNA) impairs the ability of moderately- to highly-trained female collegiate rowers to increase their training quality, as well as their performance in response to 6 weeks of iron supplementation, in addition to their usual endurance training.

This study was conducted in three phases. Phase 1 was a cross-sectional study designed to describe the iron status of a diverse sample of female collegiate rowers around central New York state. Iron status was screened with a venous blood sample, and demographic and other health and self-reported performance data were also collected. One-hundred and sixty-five female collegiate endurance athletes were screened to identify IDNA subjects (sFer <20 µg/l, Hgb >12 g/dL) for an iron supplementation trial.

Phase 2 was a cross-sectional study designed to measure and compare the metabolic and functional consequences of ID in a sample of highly-trained female rowers across a broad range of both fitness levels (novice to varsity)and iron status (normal, ID, and IDNA). This cross-sectional study was an analysis of the baseline data for potential RCT participants (IDNA) at the beginning of a training season. In addition to those IDNA subjects participating in the supplementation trial, we included a sample of non-anemic, non-iron deficient rowers. These subjects completed all baseline protocols in the lab, and recorded one week of training activities, in addition to all other baseline data collected. This cross-sectional study enabled us to investigate potential relationships between iron status and early training season performance.

This plausibility analysis was useful, in light of the putative mechanisms (correlations between iron status and physical performance), to explain how iron status may affect physical performance. These analyses suggested relationships between iron status and performance, but did not provide strong causal evidence, as temporal relationships between iron status and performance cannot be determined in a cross-sectional study. We did, however, need to identify and control confounding factors related to both iron status and performance to control bias.

Phase 3 was a randomized, placebo-controlled supplementation trial designed to explore how IDNA and iron supplementation affect iron status, performance, and training over 6-weeks of rowing training. Rowers with normal iron status were included in this study to examine training effects (if any) on iron status and performance. This study was designed to elucidate the cause-effect relationship(s) between iron status (and iron supplementation), training and performance.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking
* current member of college/university rowing team

Exclusion Criteria:

* acute or chronic injury or illness at time of screening
* physician-diagnosed asthma, musculoskeletal problems, or eating disorders
* pregnant or lactating
* use of steroids or other performance-enhancing substances

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Markers of iron status | 6 weeks

SECONDARY OUTCOMES:
Physical performance outcomes | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jere D. Haas, PhD, Principal Investigator — Cornell University; Diane M. DellaValle, PhD, Study Director — Cornell University
Locations (1):
- Human Metabolic Research Unit, MVR Hall, Cornell University, Ithaca, New York, United States

REFERENCES:
- [Result] DellaValle DM, Haas JD. Impact of iron depletion without anemia on performance in trained endurance athletes at the beginning of a training season: a study of female collegiate rowers. Int J Sport Nutr Exerc Metab. 2011 Dec;21(6):501-6. doi: 10.1123/ijsnem.21.6.501. PMID 22089308
- [Result] Dellavalle DM, Haas JD. Iron status is associated with endurance performance and training in female rowers. Med Sci Sports Exerc. 2012 Aug;44(8):1552-9. doi: 10.1249/MSS.0b013e3182517ceb. PMID 22382172
- [Result] DellaValle DM, Haas JD. Iron supplementation improves energetic efficiency in iron-depleted female rowers. Med Sci Sports Exerc. 2014 Jun;46(6):1204-15. doi: 10.1249/MSS.0000000000000208. PMID 24195864